CLINICAL TRIAL: NCT02388308
Title: Evaluation of Clarity Ultrasound Guidance for Prostate Therapy
Acronym: Clarity-Pro
Status: Completed | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 4267
Record Dates: First submitted 2015-02-20; First posted 2015-03-17 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Image-guided radiotherapy; Ultrasound guidance
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patient volunteers: Patients who have received radiotherapy for prostate cancer which included a planning CT scan, or who are currently receiving radiotherapy including a CT scan.
  Interventions: Device: Clarity ultrasound
- Gold fiducial marker group: Patients receiving radiotherapy for prostate cancer as part of a clinical trial or standard care which includes gold FM or EM insertion, or patients who have previously received RT for prostate cancer which included EM insertion.
  Interventions: Device: Clarity ultrasound
- Electromagnetic marker group: Patients receiving radiotherapy for prostate cancer as part of a clinical trial or standard care which includes gold FM or EM insertion, or patients who have previously received RT for prostate cancer which included EM insertion.
  Interventions: Device: Clarity ultrasound
- General patients: Patients who are receiving radiotherapy for prostate cancer and who are not receiving FMs. Attempts will be made to match Group 4 patients BMI and time receiving hormone therapy to patients in group 2 and 3 (see below, section 6.1 recruitment.
  Interventions: Device: Clarity ultrasound

INTERVENTIONS:
Device: Clarity ultrasound — Ultrasound imaging data will be recorded only. Treatment will not be altered as a result of this study.

SUMMARY:
Radiotherapy (RT) is an important treatment for prostate cancer with over 10,000 men receiving RT per year in the UK. Prostate RT aims to deliver radiation dose to the prostate to kill cancer cells whilst minimizing the dose given to surrounding normal tissues, such as the bladder or the rectum. Radiation is delivered in a number of daily treatments which are called 'fractions'. The position of the prostate varies each day and during the radiation delivery. To accurately aim the radiation the prostate needs to be located before daily treatment. Clarity is an ultrasound image guidance system that locates the prostate and monitors its position during treatment. Ultrasound does not give a radiation dose, is non-invasive, provides fast imaging and can easily visualise soft tissues. Before Clarity is implemented the investigators wish to ensure that it can accurately locate and monitor the prostate by comparing Clarity with marker-based techniques in 24 patients. Patients receive markers as part of other trials which are currently recruiting at The Royal Marsden (for example, patients in the DELINEATE trial and the PACE trials receive implanted gold markers and patients in the PROSPARE trial have received electromagnetic markers). Patients who have received or will be receiving markers as part of other studies will be asked to also to take part in this study. This means that there will be no additional intervention for patients as a result of this study. Clarity will be considered a safe and effective imaging system if the mean and standard deviation of the differences between Clarity measurements and marker measurements, of prostate position, are less than 1mm. It is possible that markers will influence the Clarity measurements. To find out if this happens, the mean and standard deviation of Clarity measurements in a group of 24 patients without markers to the group with markers will be compared.

Primary Aim: To evaluate the accuracy of Clarity ultrasound image guidance system for prostate motion estimation during treatment (intra-fraction), by comparison with implanted marker-based image guidance techniques.

Primary Hypothesis: Clarity can be safely used to deliver radiotherapy using similar (within 1mm) treatment margins to those that would be employed if fiducial markers based image guidance techniques were used.

ELIGIBILITY:
Inclusion Criteria:

Two patient groups and two patient volunteer groups will be recruited:

Groups 1: Patient volunteers who have received radiotherapy for prostate cancer which included a planning CT scan, or who are currently receiving radiotherapy.

Groups 2 and 3:

* Patients receiving radiotherapy for prostate cancer as part of a clinical trial or standard care which includes gold FM or EM insertion
* Patients who have previously received RT for prostate cancer which included EM insertion.

Group 4: Patients who are receiving radiotherapy for prostate cancer and who are not receiving FMs. Attempts will be made to match Group 4 patients BMI and time receiving hormone therapy to patients in group 2 and 3 (see below, section 6.1 recruitment.

Exclusion Criteria:

Groups 1 to 4: Patients who have received prostatectomy.

Groups 2 and 4: Patients receiving less than 6 RT fractions.

Group 4 only: Patients who have received FMs or EMs.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing radiotherapy for prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
Prostate position (measured in millimeters) measured using Clarity ultrasound and implanted fiducial markers | Outcome measures will be assessed for each patient during radiotherapy, an average of five weeks.
  Mean (and standard deviation) of the differences in prostate position determined using Clarity and that determined using fiducial marker based image guidance during radiotherapy delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Harris, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (1):
- The Royal Marsden, Sutton, United Kingdom

REFERENCES:
- [Derived] Grimwood A, Rivaz H, Zhou H, McNair HA, Jakubowski K, Bamber JC, Tree AC, Harris EJ. Improving 3D ultrasound prostate localisation in radiotherapy through increased automation of interfraction matching. Radiother Oncol. 2020 Aug;149:134-141. doi: 10.1016/j.radonc.2020.04.044. Epub 2020 May 6. PMID 32387546
- [Derived] Grimwood A, McNair HA, O'Shea TP, Gilroy S, Thomas K, Bamber JC, Tree AC, Harris EJ. In Vivo Validation of Elekta's Clarity Autoscan for Ultrasound-based Intrafraction Motion Estimation of the Prostate During Radiation Therapy. Int J Radiat Oncol Biol Phys. 2018 Nov 15;102(4):912-921. doi: 10.1016/j.ijrobp.2018.04.008. Epub 2018 Apr 16. PMID 29859785